CLINICAL TRIAL: NCT05683496
Title: A Phase 1/2, Adaptive, Multiple Dose Ranging Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Clinical Efficacy of Lonigutamab in Subjects With Thyroid Eye Disease (TED)
Brief Title: Efficacy and Safety of Lonigutamab in Subjects With Thyroid Eye Disease (TED)
Acronym: TED
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ACELYRIN Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 421-01-02
Record Dates: First submitted 2022-12-20; First posted 2023-01-13 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Thyroid Eye Disease
Keywords: TED
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Intervention Model Description: Up to 4 cohorts are planned, with each cohort receiving one of 5 different treatment doses
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-masked, placebo-controlled and open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Experimental): Single SC injection of dose 1 of lonigutamab or placebo at Day 1 and Day 21
  Interventions: Drug: lonigutamab; Drug: Placebo
- Cohort 2 (Experimental): multiple doses of dose 2 of lonigutamab administered SC injection weekly
  Interventions: Drug: lonigutamab
- Cohort 3 (Experimental): multiple doses of lonigutamab dose 3 administered SC injection every 4 weeks.
  Interventions: Drug: lonigutamab
- Cohort 4 (Experimental): multiple doses of lonigutamab dose 4 administered SC injection every 4 or 3 weeks.
  Interventions: Drug: lonigutamab

INTERVENTIONS:
Drug: lonigutamab — subcutaneous injection
Drug: Placebo — subcutaneous injection
  Arms: Cohort 1

SUMMARY:
Phase 1/2, multicenter, multiple dose clinical study designed to evaluate lonigutamab in subjects with TED.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, ≥18 and ≤75 years of age.
* Proptosis defined in the study eye as ≥3 mm above normal.
* Clinical Activity Score (CAS) ≥4 (using a 7-item scale) for the most severely affected eye
* Onset of active TED symptoms prior to baseline
* Must agree to use highly effective contraception as specified in the protocol

Key Exclusion Criteria:

* Pathology related to inflammatory bowel disease or irritable bowel syndrome.
* Clinically significant pathology related to hearing or history of hearing impairment
* Optic neuropathy
* Corneal decompensation unresponsive to medical management.
* Previous orbital irradiation (for any cause) or any previous surgical treatment for TED.
* Subjects with diabetes or hemoglobin A1c >6.0% at screening
* Any steroid use (intravenous [IV] or oral) with a cumulative dose equivalent to >3 g of methylprednisolone for the treatment of TED within the last year.
* Previous steroid use (IV or oral) specifically for the treatment of TED not to exceed 1 g total dose in the 8 weeks prior to Screening.
* Previous use of teprotumumab or any other IGF-1 receptor (IGF-1R) inhibitor.
* Any previous treatment with a biologic drug for the treatment of TED (eg, rituximab and tocilizumab)
* Any other immunosuppressive agent within 1 month of screening.
* Cohort 4 only: Prior history of craniofacial surgery or medical conditions that could alter orbital or facial features.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Incidence and characterization of nonserious treatment emergent adverse events (TEAEs) | Day 1 to Day 169
  Safety and Tolerability
Incidence and characterization of serious treatment emergent adverse events (TEAEs) | Day 1 to Day 169
  Safety and Tolerability

SECONDARY OUTCOMES:
PK profile of lonigutamab | Day 1 to Day 169
  minimum observed concentration (Cmin)
PK profile of lonigutamab | Day 1 to Day 169
  Maximum observed concentration (Cmax)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (6):
  - Clinical Research Site, Jacksonville, Florida
  - Clinical Research Site, Atlanta, Georgia
  - Clinical Research Site, Ann Arbor, Michigan
  - Clinical Research Site, East Setauket, New York
  - Clinical Research Site, New York, New York
  - Clinical Research Site, Morgantown, West Virginia
- Australia (5):
  - Clinical Research Site, Sydney, New South Wales
  - Clinical Research Site, Woolloongabba, Queensland
  - Clinical Research Site, Adelaide, South Australia
  - Clinical Research Site, East Melbourne, Victoria
  - Clinical Research Site, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No